CLINICAL TRIAL: NCT04745143
Title: Monotherapy of an NMDA Enhancer for Schizophrenia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMUH105-REC1-050
Record Dates: First submitted 2021-01-14; First posted 2021-02-09 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; NMDA; Oxidative stress
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NMDAE (Experimental): An NMDA enhancer
  Interventions: Drug: NMDAE
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo Cap

INTERVENTIONS:
Drug: NMDAE — Use of an NMDA enhancer for the treatment of schizophrenia
  Arms: NMDAE
Drug: Placebo Cap — Use of placebo as a comparator
  Arms: Placebo

SUMMARY:
Previous studies found that some NMDA-enhancing agent was able to augment antioxidant activity and its adjunctive therapy was better than placebo in reducing clinical symptoms and cognitive deficits and revealed favorable safety in patients with chronic schizophrenia. Of note, a substantial portion of schizophrenia patients refuse or cannot tolerate antipsychotics due to poor response or severe side effects. Therefore, this study aims to examine the efficacy and safety of an NMDA enhancer (NMDAE) as a monotherapy for the treatment of schizophrenia.

DETAILED DESCRIPTION:
Several lines of evidence suggest that schizophrenia is associated with accelerated aging and oxidative stress may play a role. Cognitive deficits are core symptoms of accelerated aging in patients with schizophrenia and the most difficult domain to treat. Current antipsychotics have limited, if any, efficacy for cognitive function. Previous studies found that some NMDA-enhancing agent was able to augment antioxidant activity and its adjunctive therapy was better than placebo in reducing not only clinical symptoms but also cognitive deficits and revealed favorable safety in patients with chronic schizophrenia. Of note, a substantial portion of schizophrenia patients refuse or cannot tolerate antipsychotics due to poor response or severe side effects. This study aims to examine the efficacy and safety of NMDAE monotherapy for the treatment of schizophrenia. The investigators enroll patients with schizophrenia who refuse or are unable to tolerate antipsychotics due to poor response or adverse effects into a 6-week randomized, double-blind trial to receive monotherapy of NMDAE or placebo. The investigators biweekly measure clinical performances and side effects. Cognitive functions are assessed at baseline and at endpoint of treatment by a battery of tests. The efficacies of NMDAE and placebo will be compared.

Chi-square (or Fisher's exact test) will be used to compare differences of categorical variables and t-test (or Mann-Whitney test if the distribution is not normal) for continuous variables between treatment groups. Mean changes from baseline in repeated-measure assessments will be assessed using the generalized estimating equation (GEE). All p values for clinical measures will be based on two-tailed tests with a significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Have a DSM-5 (American Psychiatric Association) diagnosis of schizophrenia
* Refuse or are unable to tolerate antipsychotics due to poor response or adverse effects
* PANSS total score ≥ 60
* Free of antipsychotic drugs for at least 1 week
* Agree to participate in the study and provide informed consent

Exclusion Criteria:

* Current substance abuse or history of substance dependence in the past 3 months
* History of epilepsy, head trauma, stroke or other serious medical or neurological illness which may interfere with the study
* Use of depot antipsychotic in the past 3 months;
* Clinically significant laboratory screening tests
* Pregnancy or lactation
* Inability to follow protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change of Positive and Negative Syndrome Scale (PANSS) | week 0, 2, 4, 6
  Assessment of overall symptoms. Minimum value: 30, maximum value:210, the higher scores mean a worse outcome.
Change of scales for the Assessment of Negative Symptoms (SANS) total score | week 0, 2, 4, 6
  Assessment of negative symptoms. Minimum value: 0, maximum value:100, the higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Positive subscale, Negative subscales, and General Psychopathology subscale of Positive and Negative Syndrome Scale (PANSS) | week 0, 2, 4, 6
  PANSS-positive: Assessment of positive symptoms. Minimum value: 7, maximum value:49, the higher scores mean a worse outcome.
  PANSS-negative: Assessment of negative symptoms. Minimum value: 7, maximum value:49, the higher scores mean a worse outcome.
  PANSS-general psychopathology: Assessment of general psychopathology. Minimum value: 16, maximum value:112, the higher scores mean a worse outcome.
Clinical Global Impression | week 0, 2, 4, 6
  Assessment of general impression. Minimum value: 1, maximum value:7, the higher scores mean a worse outcome.
Global Assessment of Functioning | week 0, 2, 4, 6
  Assessment of social, occupational, and psychological function. Minimum value: 1, maximum value:100, the higher scores mean better function.
Hamilton Rating Scale for Depression | week 0, 2, 4, 6
  Assessment of depressive symptoms. Minimum value: 0, maximum value:52, the higher scores mean a worse outcome.
Quality of Life Scale | week 0, 2, 4, 6
  Assessment of life quality. Minimum value: 0, maximum value:126, the higher scores mean a better outcome.
Cognitive function | Week 0, 6
  The measure is the composite from multiple measures.
  Ten cognitive tests for assessment of 7 cognitive domains:
  1. speed of processing (assessed by 3 tests: Category Fluency, Trail Marking A, WAIS-III Digit Symbol-Coding);
  2. sustained attention (Continuous Performance Test);
  3. working memory: verbal (digit span) and nonverbal (spatial span);
  4. verbal learning and memory (WMS-III, word listing);
  5. visual learning and memory (WMS-III, visual reproduction);
  6. reasoning and problem solving (WISC-III, Maze);
  7. social cognition (the Mayer-Salovey-Caruso Emotional Intelligence Test [MSCEIT] Version 2)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, China Medical University Hospital, Taichung, Taiwan